CLINICAL TRIAL: NCT04647097
Title: Recurrent Acute Pancreatitis Prevention by the Elimination of Alcohol and Cigarette Smoking (REAPPEAR): Protocol of a Randomized Controlled Trial and a Cohort Study
Brief Title: Preventing the Recurrence of Acute Pancreatitis by Alcohol and Smoking Cessation
Acronym: REAPPEAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dr Hegyi Péter, Principal Investigator, Director of the Centre for Translational Medicine at University of Pécs, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 40394-10/2020/EÜIG
Record Dates: First submitted 2020-11-16; First posted 2020-11-30 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Acute Pancreatitis; Recurrent Acute Pancreatitis
Keywords: acute pancreatitis; recurrent acute pancreatitis; smoking; alcohol; lifestyle intervention
MeSH Terms: conditions — Pancreatitis; Smoking

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial and a cohort study
Who Masked: Outcomes Assessor
Masking Description: The assessors of the outcomes will be blinded regarding allocation. The medical team providing the visits and treatment during hospitalization rwill not be aware of the allocation. Patients and the study nurse can not be blinded, due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard intervention plus repeated intervention (Active Comparator): Patients randomized to the standard intervention plus repeated intervention arm
  Interventions: Behavioral: Standard intervention plus repeated intervention
- Standard intervention only (Active Comparator): Patients randomized to the standard intervention only arm
  Interventions: Behavioral: Standard intervention only

INTERVENTIONS:
Behavioral: Standard intervention only — Standard intervention (SI) will be a part of standard care in all participating centers, and will be provided for all acute pancreatitis patients, who are hospitalized and their condition is alcohol induced. A specially trained study nurse will deliver the intervention, since they were found to be the most effective regarding the decrease in alcohol consumption and smoking. The cost- effectiveness of the intervention and the feasibility were also taken into account. The Assist-linked brief intervention according to the World Health Organization (WHO) will serve as the base for the intervention, with an avarage of 30 minutes, based on a review containing 69 randomized controlled trials, which concluded that longer intervention do not have additional benefit. The patients will be also educated about the disease course of acute pancreatitis during the standard intervention.
  Arms: Standard intervention only
Behavioral: Standard intervention plus repeated intervention — Standard intervention (SI) will be performed as described above. The repeated intervention will be delivered by the former mentioned same nurse and will be structured similarly to the standard intervention. Every visit and intervention will be individually altered according to the motivation of the patient, but they will follow the same structure. The sessions can be divided into three main parts: first, highlighting the harmful effects of smoking and alcohol on the pancreatic functions. Secondly, a discussion about the motivation of the patient will happen. The last portion of the session will focus on the responsibility of the individual to reach the desired goal will be highlighted. To enhance the efficacy of our intervention we wish to provide feed-back for the patient based on laboratory testing: the mean corpuscular volume (MCV) and gamma glutamyl-transferase (GGT) values will be measured right before the interview. The study nurse will not take part in patient care.
  Arms: Standard intervention plus repeated intervention

SUMMARY:
Recurrence of acute pancreatitis (AP) is often facilitated by regular alcohol consumption and smoking. An applied lifestyle intervention focusing on the cessation of alcohol consumption and smoking might prevent the recurrence of AP. REAPPEAR Study is a randomized controlled trial and a cohort study focusing on the efficacy of the lifestyle intervention and the effect of quitting alcohol and smoking respectively.

DETAILED DESCRIPTION:
Alcohol and smoking caused recurrent acute pancretitis might be prevented. The condition is known for it's causative effect of chronic pancreatitis and nonbeneficial effect on quality of life. Clinical equipoise regarding the impact of alcohol and smoking cessation still exists, due to the non existence of well designed clinical trials. The aim of the REAPPEAR study is to investigate the effect of cessation program of alcohol and tobacco use on the recurrence of acute pancreatitis.

The REAPPEAR Study is a combined clinical trial involving a randomized multicenter clinical trial (REAPPEAR-T), which assesses the effect of the cessation program on the recurrence of the acute pancreatitis, and a cohort analysis, which investigates the effect of smoking and alcohol cessation on the recurrance of acute pancreatitis. Daily smokers, hospitalized with alcohol-induced pancreatitis will be included in the trial. Standard cessational intervention will be provided for all patients before enrollment. Laboratory testing, measurement of blood pressure and BMI will be performed, while also hair, urine samples and blood will be retrieved for later biomarker measurement. The evaluation of motivation to change, addiction, quality of life and socioeconomic status will be recorded at every visit, which will take place every 3 months or yearly according to the random allocation. For patients, who present at visit of every 3 months a brief intervention will be provided, together with a laboratory testing to provide feedback. The primary composite endpoint of this study will be the recurrence rate of acute pancreatitis irrespective of etiology and all-cause mortality in a 2 year timeframe. The cost-effectiveness will be also evaluated.

ELIGIBILITY:
Inclusion criteria:

* Patient hospitalized with alcohol-induced AP (defined by the revised Atlanta criteria 38)
* Every day smoker (defined as an adult patient who smoked at least 100 cigarettes in his or her lifetime, and now smokes on a daily basis; as per the CDC definition), with at least 1-year history of smoking
* Aged 18-80 years
* Provided written informed consent
* Willing to participate in the intervention in every three months

Exclusion criteria:

* Possible etiologies for AP other than alcohol (eg. gallstone-related, hypertriglyceridemia above 11.5 mM 40-42, hypercalcemia, viral infection) if the etiological cannot be terminated during the index admission (lack of same admission cholecystectomy, familiar hypertrygliceridemia) and cases with combined etiological factors will be excluded
* Untreated, decompensated or severe mMajor psychiatric illnesses (e.g. schizophrenia, bipolar disorder, dementia)
* Currently taking part in a smoking cessation program
* Undergoing active or palliative treatment for malignancy
* Pregnancy, breastfeeding
* Life expectancy is less than two years
* Didn't agreed to participate
* Other

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of recurrence rate of AP and all cause mortality | 24 months
  Recurrence rate of AP irrespective of etiology and all cause mortality. The diagnosis of AP based on the two out of three rule. (At least 2 of 3 typical features are present -upper abdominal pain, elevation of serum pancreatic enzymes at least 3 times the reference value, and imaging findings consistent with AP.)

SECONDARY OUTCOMES:
Recurrence of acute pancreatitis irrespective of etiology | 6, 18,24 months
  Recurrence of acute pancreatitis irrespective of etiology given as cumulative incidence and as rate of event
Recurrence of alcohol-induced AP | 24 months
  Recurrence of alcohol-induced AP given as rate of event
Likely pancreatitis | 3, 6, 9, 12, 15, 18, 21, 24 months
  Likely pancreatitis, fulfilling the diagnostic criteria of epigastric pain, a serum amylase or lipase level at least two times the upper normal level, and elevated leukocyte count or CRP levels
Length of hospital stay | 3, 6, 9, 12, 15, 18, 21, 24 months
  Length of hospital stay given in days due to recurrent pancreatitis and overall during follow-up
Presentation to the emergency unit, hospital re-admission | 3, 6, 9, 12, 15, 18, 21, 24 months
  Presentation to the emergency unit, hospital re-admission given as cumulative incidence
Development of chronic pancreatitis | 3, 6, 9, 12, 15, 18, 21, 24 months
  Development of chronic pancreatitis given as incidence within 2 years
Healthcare cost | 3, 6, 9, 12, 15, 18, 21, 24 months
  Healthcare cost from the perspective of the health insurance fund within 2 years
Quality adjusted life years | 3, 6, 9, 12, 15, 18, 21, 24 months
  Quality adjusted life years (QALY) within 2 year
Change of alcohol consumption given in gram per week | 3, 6, 9, 12, 15, 18, 21, 24 months
  Change of alcohol consumption compared to baseline given in gram per week based on patient reported data
Change of tobacco use given in pieces per day | 3, 6, 9, 12, 15, 18, 21, 24 months
  Change of tobacco use compared to the baseline given in pieces per day based on patient reported data
Change of alcohol consumption | 3, 6, 9, 12, 15, 18, 21, 24 months
  Change of alcohol consumption compared to baseline estimated from biomarker levels

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Translational Medicine, University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wadhwa V, Patwardhan S, Garg SK, Jobanputra Y, Lopez R, Sanaka MR. Health Care Utilization and Costs Associated With Acute Pancreatitis. Pancreas. 2017 Mar;46(3):410-415. doi: 10.1097/MPA.0000000000000755. PMID 28099261
- [Background] Szentesi A, Toth E, Balint E, Fanczal J, Madacsy T, Laczko D, Ignath I, Balazs A, Pallagi P, Maleth J, Rakonczay Z Jr, Kui B, Illes D, Marta K, Blasko A, Demcsak A, Parniczky A, Par G, Godi S, Mosztbacher D, Szucs A, Halasz A, Izbeki F, Farkas N, Hegyi P; Hungarian Pancreatic Study Group. Analysis of Research Activity in Gastroenterology: Pancreatitis Is in Real Danger. PLoS One. 2016 Oct 24;11(10):e0165244. doi: 10.1371/journal.pone.0165244. eCollection 2016. PMID 27776171
- [Background] Machicado JD, Yadav D. Epidemiology of Recurrent Acute and Chronic Pancreatitis: Similarities and Differences. Dig Dis Sci. 2017 Jul;62(7):1683-1691. doi: 10.1007/s10620-017-4510-5. Epub 2017 Mar 9. PMID 28281168
- [Background] Tenner S, Baillie J, DeWitt J, Vege SS; American College of Gastroenterology. American College of Gastroenterology guideline: management of acute pancreatitis. Am J Gastroenterol. 2013 Sep;108(9):1400-15; 1416. doi: 10.1038/ajg.2013.218. Epub 2013 Jul 30. PMID 23896955
- [Background] Guda NM, Muddana V, Whitcomb DC, Levy P, Garg P, Cote G, Uc A, Varadarajulu S, Vege SS, Chari ST, Forsmark CE, Yadav D, Reddy DN, Tenner S, Johnson CD, Akisik F, Saluja AK, Lerch MM, Mallery JS, Freeman ML. Recurrent Acute Pancreatitis: International State-of-the-Science Conference With Recommendations. Pancreas. 2018 Jul;47(6):653-666. doi: 10.1097/MPA.0000000000001053. PMID 29894415
- [Background] Yadav D, O'Connell M, Papachristou GI. Natural history following the first attack of acute pancreatitis. Am J Gastroenterol. 2012 Jul;107(7):1096-103. doi: 10.1038/ajg.2012.126. Epub 2012 May 22. PMID 22613906
- [Background] Cote GA, Yadav D, Abberbock JA, Whitcomb DC, Sherman S, Sandhu BS, Anderson MA, Lewis MD, Alkaade S, Singh VK, Baillie J, Banks PA, Conwell D, Guda NM, Muniraj T, Tang G, Brand R, Gelrud A, Amann ST, Forsmark CE, Wilcox MC, Slivka A, Gardner TB. Recurrent Acute Pancreatitis Significantly Reduces Quality of Life Even in the Absence of Overt Chronic Pancreatitis. Am J Gastroenterol. 2018 Jun;113(6):906-912. doi: 10.1038/s41395-018-0087-7. Epub 2018 Jun 5. PMID 29867178
- [Background] Mandalia A, Wamsteker EJ, DiMagno MJ. Recent advances in understanding and managing acute pancreatitis. F1000Res. 2018 Jun 28;7:F1000 Faculty Rev-959. doi: 10.12688/f1000research.14244.2. eCollection 2018. PMID 30026919
- [Background] Krishna SG, Kamboj AK, Hart PA, Hinton A, Conwell DL. The Changing Epidemiology of Acute Pancreatitis Hospitalizations: A Decade of Trends and the Impact of Chronic Pancreatitis. Pancreas. 2017 Apr;46(4):482-488. doi: 10.1097/MPA.0000000000000783. PMID 28196021
- [Background] Nikkola J, Raty S, Laukkarinen J, Seppanen H, Lappalainen-Lehto R, Jarvinen S, Nordback I, Sand J. Abstinence after first acute alcohol-associated pancreatitis protects against recurrent pancreatitis and minimizes the risk of pancreatic dysfunction. Alcohol Alcohol. 2013 Jul-Aug;48(4):483-6. doi: 10.1093/alcalc/agt019. Epub 2013 Mar 28. PMID 23538610
- [Background] Magnusdottir BA, Baldursdottir MB, Kalaitzakis E, Bjornsson ES. Risk factors for chronic and recurrent pancreatitis after first attack of acute pancreatitis. Scand J Gastroenterol. 2019 Jan;54(1):87-94. doi: 10.1080/00365521.2018.1550670. Epub 2019 Jan 31. PMID 30700163
- [Background] Nikkola J, Laukkarinen J, Lahtela J, Seppanen H, Jarvinen S, Nordback I, Sand J. The Long-term Prospective Follow-up of Pancreatic Function After the First Episode of Acute Alcoholic Pancreatitis: Recurrence Predisposes One to Pancreatic Dysfunction and Pancreatogenic Diabetes. J Clin Gastroenterol. 2017 Feb;51(2):183-190. doi: 10.1097/MCG.0000000000000564. PMID 28060789
- [Background] Nordback I, Pelli H, Lappalainen-Lehto R, Jarvinen S, Raty S, Sand J. The recurrence of acute alcohol-associated pancreatitis can be reduced: a randomized controlled trial. Gastroenterology. 2009 Mar;136(3):848-55. doi: 10.1053/j.gastro.2008.11.044. Epub 2008 Nov 27. PMID 19162029
- [Background] Lappalainen-Lehto R, Koistinen N, Aalto M, Huhtala H, Sand J, Nordback I, Seppa K. Goal-related outcome after acute alcohol-pancreatitis -- a two-year follow-up study. Addict Behav. 2013 Dec;38(12):2805-9. doi: 10.1016/j.addbeh.2013.07.008. Epub 2013 Jul 21. PMID 24018221
- [Background] Tolstrup JS, Kristiansen L, Becker U, Gronbaek M. Smoking and risk of acute and chronic pancreatitis among women and men: a population-based cohort study. Arch Intern Med. 2009 Mar 23;169(6):603-9. doi: 10.1001/archinternmed.2008.601. PMID 19307524
- [Background] Lindkvist B, Appelros S, Regner S, Manjer J. A prospective cohort study on risk of acute pancreatitis related to serum triglycerides, cholesterol and fasting glucose. Pancreatology. 2012 Jul-Aug;12(4):317-24. doi: 10.1016/j.pan.2012.05.002. Epub 2012 May 10. PMID 22898632
- [Background] Sadr-Azodi O, Andren-Sandberg A, Orsini N, Wolk A. Cigarette smoking, smoking cessation and acute pancreatitis: a prospective population-based study. Gut. 2012 Feb;61(2):262-7. doi: 10.1136/gutjnl-2011-300566. Epub 2011 Aug 11. PMID 21836026
- [Background] Majumder S, Gierisch JM, Bastian LA. The association of smoking and acute pancreatitis: a systematic review and meta-analysis. Pancreas. 2015 May;44(4):540-6. doi: 10.1097/MPA.0000000000000301. PMID 25872130
- [Background] Schuckit MA. Alcohol-use disorders. Lancet. 2009 Feb 7;373(9662):492-501. doi: 10.1016/S0140-6736(09)60009-X. Epub 2009 Jan 23. PMID 19168210
- [Background] Peris P, Pares A, Guanabens N, Del Rio L, Pons F, Martinez de Osaba MJ, Monegal A, Caballeria J, Rodes J, Munoz-Gomez J. Bone mass improves in alcoholics after 2 years of abstinence. J Bone Miner Res. 1994 Oct;9(10):1607-12. doi: 10.1002/jbmr.5650091014. PMID 7817807
- [Background] Aguilera MT, de la Sierra A, Coca A, Estruch R, Fernandez-Sola J, Urbano-Marquez A. Effect of alcohol abstinence on blood pressure: assessment by 24-hour ambulatory blood pressure monitoring. Hypertension. 1999 Feb;33(2):653-7. doi: 10.1161/01.hyp.33.2.653. PMID 10024322
- [Background] Seitz HK, Bataller R, Cortez-Pinto H, Gao B, Gual A, Lackner C, Mathurin P, Mueller S, Szabo G, Tsukamoto H. Alcoholic liver disease. Nat Rev Dis Primers. 2018 Aug 16;4(1):16. doi: 10.1038/s41572-018-0014-7. PMID 30115921
- [Background] Jandikova H, Duskova M, Starka L. The influence of smoking and cessation on the human reproductive hormonal balance. Physiol Res. 2017 Sep 26;66(Suppl 3):S323-S331. doi: 10.33549/physiolres.933724. PMID 28948816
- [Background] Taylor DH Jr, Hasselblad V, Henley SJ, Thun MJ, Sloan FA. Benefits of smoking cessation for longevity. Am J Public Health. 2002 Jun;92(6):990-6. doi: 10.2105/ajph.92.6.990. PMID 12036794
- [Background] Parniczky A, Kui B, Szentesi A, Balazs A, Szucs A, Mosztbacher D, Czimmer J, Sarlos P, Bajor J, Godi S, Vincze A, Illes A, Szabo I, Par G, Takacs T, Czako L, Szepes Z, Rakonczay Z, Izbeki F, Gervain J, Halasz A, Novak J, Crai S, Hritz I, Gog C, Sumegi J, Golovics P, Varga M, Bod B, Hamvas J, Varga-Muller M, Papp Z, Sahin-Toth M, Hegyi P; Hungarian Pancreatic Study Group. Prospective, Multicentre, Nationwide Clinical Data from 600 Cases of Acute Pancreatitis. PLoS One. 2016 Oct 31;11(10):e0165309. doi: 10.1371/journal.pone.0165309. eCollection 2016. PMID 27798670
- [Background] Szucs A, Marjai T, Szentesi A, Farkas N, Parniczky A, Nagy G, Kui B, Takacs T, Czako L, Szepes Z, Nemeth BC, Vincze A, Par G, Szabo I, Sarlos P, Illes A, Godi S, Izbeki F, Gervain J, Halasz A, Farkas G, Leindler L, Kelemen D, Papp R, Szmola R, Varga M, Hamvas J, Novak J, Bod B, Sahin-Toth M, Hegyi P; Hungarian Pancreatic Study Group. Chronic pancreatitis: Multicentre prospective data collection and analysis by the Hungarian Pancreatic Study Group. PLoS One. 2017 Feb 16;12(2):e0171420. doi: 10.1371/journal.pone.0171420. eCollection 2017. PMID 28207747
- [Background] Yardley MM, Mirbaba MM, Ray LA. Pharmacological Options for Smoking Cessation in Heavy-Drinking Smokers. CNS Drugs. 2015;29(10):833-45. doi: 10.1007/s40263-015-0284-5. PMID 26507831
- [Background] Weinberger AH, Platt J, Jiang B, Goodwin RD. Cigarette Smoking and Risk of Alcohol Use Relapse Among Adults in Recovery from Alcohol Use Disorders. Alcohol Clin Exp Res. 2015 Oct;39(10):1989-96. doi: 10.1111/acer.12840. Epub 2015 Sep 13. PMID 26365044
- [Background] Mirbaba M. Heavy-Drinking Smokers: Pathophysiology and Pharmacologic Treatment Options. American Journal of Psychiatry Residents' Journal. 2016;11(6):8-11.
- [Background] Fucito LM, Hanrahan TH. Heavy-Drinking Smokers' Treatment Needs and Preferences: A Mixed-Methods Study. J Subst Abuse Treat. 2015 Dec;59:38-44. doi: 10.1016/j.jsat.2015.07.001. Epub 2015 Jul 14. PMID 26297324
- [Background] McKelvey K, Thrul J, Ramo D. Impact of quitting smoking and smoking cessation treatment on substance use outcomes: An updated and narrative review. Addict Behav. 2017 Feb;65:161-170. doi: 10.1016/j.addbeh.2016.10.012. Epub 2016 Oct 27. PMID 27816663
- [Background] Toll BA, Martino S, O'Malley SS, Fucito LM, McKee SA, Kahler CW, Rojewski AM, Mahoney MC, Wu R, Celestino P, Seshadri S, Koutsky J, Hyland A, Cummings KM. A randomized trial for hazardous drinking and smoking cessation for callers to a quitline. J Consult Clin Psychol. 2015 Jun;83(3):445-54. doi: 10.1037/a0038183. Epub 2014 Nov 24. PMID 25419583
- [Background] Crockett SD, Wani S, Gardner TB, Falck-Ytter Y, Barkun AN; American Gastroenterological Association Institute Clinical Guidelines Committee. American Gastroenterological Association Institute Guideline on Initial Management of Acute Pancreatitis. Gastroenterology. 2018 Mar;154(4):1096-1101. doi: 10.1053/j.gastro.2018.01.032. Epub 2018 Feb 3. No abstract available. PMID 29409760
- [Background] Working Group IAP/APA Acute Pancreatitis Guidelines. IAP/APA evidence-based guidelines for the management of acute pancreatitis. Pancreatology. 2013 Jul-Aug;13(4 Suppl 2):e1-15. doi: 10.1016/j.pan.2013.07.063. PMID 24054878
- [Background] Samarasekera E, Mahammed S, Carlisle S, Charnley R; Guideline Committee. Pancreatitis: summary of NICE guidance. BMJ. 2018 Sep 5;362:k3443. doi: 10.1136/bmj.k3443. No abstract available. PMID 30185473
- [Background] Isaji S, Takada T, Mayumi T, Yoshida M, Wada K, Yokoe M, Itoi T, Gabata T. Revised Japanese guidelines for the management of acute pancreatitis 2015: revised concepts and updated points. J Hepatobiliary Pancreat Sci. 2015 Jun;22(6):433-45. doi: 10.1002/jhbp.260. PMID 25904407
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Yadav D. Reassessing the Risk of Pancreatitis With Alcohol. Pancreas. 2016 Jul;45(6):781-2. doi: 10.1097/MPA.0000000000000668. No abstract available. PMID 27295528
- [Background] Mosztbacher D, Hanak L, Farkas N, Szentesi A, Miko A, Bajor J, Sarlos P, Czimmer J, Vincze A, Hegyi PJ, Eross B, Takacs T, Czako L, Nemeth BC, Izbeki F, Halasz A, Gajdan L, Hamvas J, Papp M, Foldi I, Feher KE, Varga M, Csefko K, Torok I, Farkas HP, Mickevicius A, Maldonado ER, Sallinen V, Novak J, Ince AT, Galeev S, Bod B, Sumegi J, Pencik P, Dubravcsik Z, Illes D, Godi S, Kui B, Marta K, Pecsi D, Varju P, Szakacs Z, Darvasi E, Parniczky A, Hegyi P; Hungarian Pancreatic Study Group. Hypertriglyceridemia-induced acute pancreatitis: A prospective, multicenter, international cohort analysis of 716 acute pancreatitis cases. Pancreatology. 2020 Jun;20(4):608-616. doi: 10.1016/j.pan.2020.03.018. Epub 2020 Apr 10. PMID 32402696
- [Background] Zadori N, Gede N, Antal J, Szentesi A, Alizadeh H, Vincze A, Izbeki F, Papp M, Czako L, Varga M, de-Madaria E, Petersen OH, Singh VP, Mayerle J, Faluhelyi N, Miseta A, Reiber I, Hegyi P. EarLy Elimination of Fatty Acids iN hypertriglyceridemia-induced acuTe pancreatitis (ELEFANT trial): Protocol of an open-label, multicenter, adaptive randomized clinical trial. Pancreatology. 2020 Apr;20(3):369-376. doi: 10.1016/j.pan.2019.12.018. Epub 2019 Dec 30. PMID 31959416
- [Background] Szentesi A, Parniczky A, Vincze A, Bajor J, Godi S, Sarlos P, Gede N, Izbeki F, Halasz A, Marta K, Dobszai D, Torok I, Farkas H, Papp M, Varga M, Hamvas J, Novak J, Mickevicius A, Maldonado ER, Sallinen V, Illes D, Kui B, Eross B, Czako L, Takacs T, Hegyi P. Multiple Hits in Acute Pancreatitis: Components of Metabolic Syndrome Synergize Each Other's Deteriorating Effects. Front Physiol. 2019 Sep 20;10:1202. doi: 10.3389/fphys.2019.01202. eCollection 2019. PMID 31620021
- [Background] Hegyi P, Erőss B, Mátrai P, Hamvas J, Pécsi D, Németh B, et al. The first definition for early chronic pancreatitis. Pancreatology. 2018;18(4, Supplement):S172.
- [Background] Lohr JM, Dominguez-Munoz E, Rosendahl J, Besselink M, Mayerle J, Lerch MM, Haas S, Akisik F, Kartalis N, Iglesias-Garcia J, Keller J, Boermeester M, Werner J, Dumonceau JM, Fockens P, Drewes A, Ceyhan G, Lindkvist B, Drenth J, Ewald N, Hardt P, de Madaria E, Witt H, Schneider A, Manfredi R, Brondum FJ, Rudolf S, Bollen T, Bruno M; HaPanEU/UEG Working Group. United European Gastroenterology evidence-based guidelines for the diagnosis and therapy of chronic pancreatitis (HaPanEU). United European Gastroenterol J. 2017 Mar;5(2):153-199. doi: 10.1177/2050640616684695. Epub 2017 Jan 16. PMID 28344786
- [Background] Platt L, Melendez-Torres GJ, O'Donnell A, Bradley J, Newbury-Birch D, Kaner E, Ashton C. How effective are brief interventions in reducing alcohol consumption: do the setting, practitioner group and content matter? Findings from a systematic review and metaregression analysis. BMJ Open. 2016 Aug 11;6(8):e011473. doi: 10.1136/bmjopen-2016-011473. PMID 27515753
- [Background] Demetriou AA, Brown RS Jr, Busuttil RW, Fair J, McGuire BM, Rosenthal P, Am Esch JS 2nd, Lerut J, Nyberg SL, Salizzoni M, Fagan EA, de Hemptinne B, Broelsch CE, Muraca M, Salmeron JM, Rabkin JM, Metselaar HJ, Pratt D, De La Mata M, McChesney LP, Everson GT, Lavin PT, Stevens AC, Pitkin Z, Solomon BA. Prospective, randomized, multicenter, controlled trial of a bioartificial liver in treating acute liver failure. Ann Surg. 2004 May;239(5):660-7; discussion 667-70. doi: 10.1097/01.sla.0000124298.74199.e5. PMID 15082970
- [Background] WHO ASSIST Working Group. The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): development, reliability and feasibility. Addiction. 2002 Sep;97(9):1183-94. doi: 10.1046/j.1360-0443.2002.00185.x. PMID 12199834
- [Background] Kaner EF, Beyer FR, Muirhead C, Campbell F, Pienaar ED, Bertholet N, Daeppen JB, Saunders JB, Burnand B. Effectiveness of brief alcohol interventions in primary care populations. Cochrane Database Syst Rev. 2018 Feb 24;2(2):CD004148. doi: 10.1002/14651858.CD004148.pub4. PMID 29476653
- [Background] Kristenson H, Ohlin H, Hulten-Nosslin MB, Trell E, Hood B. Identification and intervention of heavy drinking in middle-aged men: results and follow-up of 24-60 months of long-term study with randomized controls. Alcohol Clin Exp Res. 1983 Spring;7(2):203-9. doi: 10.1111/j.1530-0277.1983.tb05441.x. PMID 6135365
- [Background] Pelli H, Lappalainen-Lehto R, Piironen A, Sand J, Nordback I. Risk factors for recurrent acute alcohol-associated pancreatitis: a prospective analysis. Scand J Gastroenterol. 2008;43(5):614-21. doi: 10.1080/00365520701843027. PMID 18415757
- [Background] Kim S, Apelberg BJ, Avila-Tang E, Hepp L, Yun D, Samet JM, Breysse PN. Utility and cutoff value of hair nicotine as a biomarker of long-term tobacco smoke exposure, compared to salivary cotinine. Int J Environ Res Public Health. 2014 Aug 15;11(8):8368-82. doi: 10.3390/ijerph110808368. PMID 25153466
- [Background] Andresen-Streichert H, Muller A, Glahn A, Skopp G, Sterneck M. Alcohol Biomarkers in Clinical and Forensic Contexts. Dtsch Arztebl Int. 2018 May 4;115(18):309-315. doi: 10.3238/arztebl.2018.0309. PMID 29807559
- [Background] Miko A, Eross B, Sarlos P, Hegyi P Jr, Marta K, Pecsi D, Vincze A, Bodis B, Nemes O, Faluhelyi N, Farkas O, Papp R, Kelemen D, Szentesi A, Hegyi E, Papp M, Czako L, Izbeki F, Gajdan L, Novak J, Sahin-Toth M, Lerch MM, Neoptolemos J, Petersen OH, Hegyi P. Observational longitudinal multicentre investigation of acute pancreatitis (GOULASH PLUS): follow-up of the GOULASH study, protocol. BMJ Open. 2019 Sep 3;9(8):e025500. doi: 10.1136/bmjopen-2018-025500. PMID 31481363
- [Background] Marta K, Szabo AN, Pecsi D, Varju P, Bajor J, Godi S, Sarlos P, Miko A, Szemes K, Papp M, Tornai T, Vincze A, Marton Z, Vincze PA, Lanko E, Szentesi A, Molnar T, Hagendorn R, Faluhelyi N, Battyani I, Kelemen D, Papp R, Miseta A, Verzar Z, Lerch MM, Neoptolemos JP, Sahin-Toth M, Petersen OH, Hegyi P; Hungarian Pancreatic Study Group. High versus low energy administration in the early phase of acute pancreatitis (GOULASH trial): protocol of a multicentre randomised double-blind clinical trial. BMJ Open. 2017 Sep 14;7(9):e015874. doi: 10.1136/bmjopen-2017-015874. PMID 28912191
- [Background] Parniczky A, Mosztbacher D, Zsoldos F, Toth A, Lasztity N, Hegyi P; Hungarian Pancreatic Study Group and the International Association of Pancreatology. Analysis of Pediatric Pancreatitis (APPLE Trial): Pre-Study Protocol of a Multinational Prospective Clinical Trial. Digestion. 2016;93(2):105-10. doi: 10.1159/000441353. Epub 2015 Nov 26. PMID 26613586
- [Background] Parniczky A, Abu-El-Haija M, Husain S, Lowe M, Oracz G, Sahin-Toth M, Szabo FK, Uc A, Wilschanski M, Witt H, Czako L, Grammatikopoulos T, Rasmussen IC, Sutton R, Hegyi P. EPC/HPSG evidence-based guidelines for the management of pediatric pancreatitis. Pancreatology. 2018 Mar;18(2):146-160. doi: 10.1016/j.pan.2018.01.001. Epub 2018 Jan 4. PMID 29398347
- [Background] Hritz I, Czako L, Dubravcsik Z, Farkas G, Kelemen D, Lasztity N, Morvay Z, Olah A, Pap A, Parniczky A, Sahin-Toth M, Szentkereszti Z, Szmola R, Szucs A, Takacs T, Tiszlavicz L, Hegyi P; Magyar Hasnyalmirigy Munkacsoport, Hungarian Pancreatic Study Group. [Acute pancreatitis. Evidence-based practice guidelines, prepared by the Hungarian Pancreatic Study Group]. Orv Hetil. 2015 Feb 15;156(7):244-61. doi: 10.1556/OH.2015.30059. Hungarian. PMID 25661970
- [Background] Gholam PM. Prognosis and Prognostic Scoring Models for Alcoholic Liver Disease and Acute Alcoholic Hepatitis. Clin Liver Dis. 2016 Aug;20(3):491-7. doi: 10.1016/j.cld.2016.02.007. Epub 2016 May 14. PMID 27373611
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Varga L. Segítségnyújtás kockázatos ivók számára National Addiction Institute; 2006.
- [Background] Németh ZK, Urbán, Róbert, Farkas, Judit, Kuntsche, Emmanuel, Demetrovics, Zsolt. Hungarian adaptation of the long and the short form of the drinking motives questionnaire (DMQ-R). Magyar Pszichológiai Szemle, 67 (4) pp 673-694. 2012.
- [Background] Kuntsche E, Kuntsche S. Development and validation of the Drinking Motive Questionnaire Revised Short Form (DMQ-R SF). J Clin Child Adolesc Psychol. 2009 Nov;38(6):899-908. doi: 10.1080/15374410903258967. PMID 20183672
- [Background] Hedman L, Katsaounou PA, Filippidis FT, Ravara SB, Lindberg A, Janson C, Gratziou C, Rohde G, Kyriakos CN, Mons U, Fernandez E, Trofor AC, Demjen T, Przewozniak K, Tountas Y, Fong GT, Vardavas CI; EUREST-PLUS consortium. Receiving support to quit smoking and quit attempts among smokers with and without smoking related diseases: Findings from the EUREST-PLUS ITC Europe Surveys. Tob Induc Dis. 2019 Mar 20;16:A14. doi: 10.18332/tid/102787. eCollection 2018. PMID 31516468
- [Background] Rencz F, Gulacsi L, Drummond M, Golicki D, Prevolnik Rupel V, Simon J, Stolk EA, Brodszky V, Baji P, Zavada J, Petrova G, Rotar A, Pentek M. EQ-5D in Central and Eastern Europe: 2000-2015. Qual Life Res. 2016 Nov;25(11):2693-2710. doi: 10.1007/s11136-016-1375-6. Epub 2016 Jul 29. PMID 27472992
- [Background] Lloyd A, Pickard AS. The EQ-5D and the EuroQol Group. Value Health. 2019 Jan;22(1):21-22. doi: 10.1016/j.jval.2018.12.002. No abstract available. PMID 30661629
- [Background] Koncz B, Darvasi E, Erdosi D, Szentesi A, Marta K, Eross B, Pecsi D, Gyongyi Z, Giran J, Farkas N, Papp M, Feher E, Vitalis Z, Janka T, Vincze A, Izbeki F, Dunas-Varga V, Gajdan L, Torok I, Karoly S, Antal J, Zadori N, Lerch MM, Neoptolemos J, Sahin-Toth M, Petersen OH, Hegyi P. LIFEStyle, Prevention and Risk of Acute PaNcreatitis (LIFESPAN): protocol of a multicentre and multinational observational case-control study. BMJ Open. 2020 Jan 6;10(1):e029660. doi: 10.1136/bmjopen-2019-029660. PMID 31911510
- [Background] Younge JO, Kouwenhoven-Pasmooij TA, Freak-Poli R, Roos-Hesselink JW, Hunink MM. Randomized study designs for lifestyle interventions: a tutorial. Int J Epidemiol. 2015 Dec;44(6):2006-19. doi: 10.1093/ije/dyv183. Epub 2015 Sep 15. PMID 26377509
- [Background] Sheron N. Alcohol and liver disease in Europe--Simple measures have the potential to prevent tens of thousands of premature deaths. J Hepatol. 2016 Apr;64(4):957-67. doi: 10.1016/j.jhep.2015.11.006. Epub 2015 Nov 16. PMID 26592352
- [Background] Sahin-Toth M, Hegyi P. Smoking and Drinking Synergize in Pancreatitis: Multiple Hits on Multiple Targets. Gastroenterology. 2017 Dec;153(6):1479-1481. doi: 10.1053/j.gastro.2017.10.031. Epub 2017 Oct 31. No abstract available. PMID 29100845
- [Derived] Ocskay K, Juhasz MF, Farkas N, Zadori N, Szako L, Szakacs Z, Szentesi A, Eross B, Miklos E, Zemplenyi A, Birkas B, Csatho A, Hartung I, Nagy T, Czopf L, Izbeki F, Gajdan L, Papp M, Czako L, Illes D, Marino MV, Mirabella A, Malecka-Panas E, Zatorski H, Susak Y, Opalchuk K, Capurso G, Apadula L, Gheorghe C, Saizu IA, Petersen OH, de-Madaria E, Rosendahl J, Parniczky A, Hegyi P; Hungarian Pancreatic Study Group. Recurrent acute pancreatitis prevention by the elimination of alcohol and cigarette smoking (REAPPEAR): protocol of a randomised controlled trial and a cohort study. BMJ Open. 2022 Jan 4;12(1):e050821. doi: 10.1136/bmjopen-2021-050821. PMID 34983758
- See also: Capacities HMoH. Az Emberi Erőforrások Minisztériuma egészségügyi szakmai irányelve a dohányzásról való leszokás támogatásáról. https://tudogyogyasz.hu2019. — https://tudogyogyasz.hu/Media/Download/12698